CLINICAL TRIAL: NCT02104804
Title: A Multicenter, Randomized, Double-Blind, Phase 3b Trial to Evaluate the Efficacy and Safety of Saxagliptin Added to Insulin Monotherapy or to Insulin in Combination With Metformin in Chinese Subjects in China With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Insulin Alone or on Insulin in Combination With Metformin
Brief Title: Evaluate the Efficacy and Safety of Saxagliptin Added to Insulin Monotherapy or to Insulin Combined With Metformin in Chinese Subjects With Type 2 Diabetes Who Have Inadequate Glycaemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00010; 2014L00001 (Other: China: State Food and Drug Administration)
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus, Insulin, Dipeptidyl-Peptidase 4 Inhibitors, Metformin,saxagliptin,Endocrine System Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — saxagliptin; Insulin, Short-Acting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saxagliptin 5mg (Experimental): Saxagliptin 5mg, administered to subjects with Type 2 diabetes inadequately controlled with insulin alone or with insulin plus metformin
  Interventions: Drug: Saxagliptin 5mg
- Placebo (Placebo Comparator): Placebo administered to subjects with Type 2 diabetes inadequately controlled with insulin alone or with insulin plus metformin
  Interventions: Drug: Placebo for Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin 5mg — Saxagliptin 5mg (plus stable insulin dose), given orally once daily (24 weeks); subjects stratified by use of stable metformin dose; flexible insulin dose (as needed for rescue).
  Other Names: Insulin: intermediate-acting or basal or premixed ( include short- or rapid-acting insulin as one component). ≥20 unit/day, ≤150 units/day; Metformin: Glucophage, 500-2500mg/day
  Arms: Saxagliptin 5mg
Drug: Placebo for Saxagliptin — Placebo tablets (plus stable insulin dose), given orally once daily (24 weeks); subjects stratified by use of stable metformin dose; flexible insulin dose (as needed for rescue).
  Other Names: Insulin: intermediate-acting or basal or premixed ( include short- or rapid-acting insulin as one component). ≥20 unit/day, ≤150 units/day; Metformin: Glucophage, 500-2500mg/day
  Arms: Placebo

SUMMARY:
A Multicenter, Randomized, Double-Blind, Phase 3b Trial to Evaluate the Efficacy and Safety of Saxagliptin Added to Insulin Monotherapy or to Insulin in Combination with Metformin in Chinese Subjects in China with Type 2 Diabetes Who Have Inadequate Glycaemic Control on Insulin Alone or on Insulin in Combination with Metformin

DETAILED DESCRIPTION:
Study Design: Randomized, prospective, double-blind, two-arm, parallel group, multi-center trial.

Target Subject Population: Subjects aged ≥18 who have type 2 diabetes (HbA1c of ≥7.5% and ≤11.0% and FPG<270 mg/dL (15 mmol/L)) on stable baseline therapy (insulin alone or insulin combined with metformin, with insulin at doses of ≥20 and ≤150 units per day total) for at least eight weeks at the time of screening. Insulin may be long-acting, intermediate-acting, or pre-mixed. 444 patients are planned to be randomized.

Investigational Product, Dosage and Mode of administration: Active treatment will comprise Saxagliptin 5 mg tablets once daily.

Comparator, Dosage and Mode of administration: Matching placebo tablets will be used as comparator.

Duration of Treatment: The study is divided to a single blind placebo lead in period of 8 weeks and a double-blind treatment phase of 24 weeks. Patients will be rescued based on high FPG values.

Statistical Methods: The analysis of the primary endpoint of change from baseline to week 24 of treatment in HbA1c will consist of an analysis of covariance (ANCOVA) model with treatment group and metformin use at enrolment as fixed effects and baseline HbA1c value as a covariate. The analysis will be performed on the Full analysis Set (FAS) consisting of randomised subjects who received at least 1 randomised investigational product dose and had at least 1 non-missing baseline and 1 post-baseline efficacy assessment. Within the framework of the ANCOVA model, point estimates and two-sided 95% confidence intervals (CI) for the mean change within each treatment group as well as for the difference in mean change between treatment groups will be calculated.

The Per Protocol (PP) analysis set is a subset of the full analysis set and will consist of subjects who do not deviate from the terms of the protocol which may affect the study outcome significantly as specified in the pre-defined protocol deviation list prior to unblinding the study. All decisions to exclude subjects from the primary data set will be made prior to the unblinding of the study. The primary efficacy endpoint of change from baseline in HbA1c, demographics, and baseline diabetes related characteristics and all secondary efficacy endpoints are to be analyzed using the PP Data Set. The analyses of PPG AUC, 120 minute PPG, FPG and mean total daily dose of insulin will also be done on the FAS and use a similar ANCOVA model as described above. Subjects achieving a therapeutic glycaemic response (A1C <7%) will be analyzed using a Fisher's exact test and will include exact 95% confidence intervals. The FPG analyses will utilize the mean of the latest two FPG values prior to randomization as the baseline value. The endpoint for the FPG analysis will be the mean of the week 20 and week 24 FPG values. All analyses (except the analysis of mean total daily dose of insulin) will utilize only observations at visits prior to rescue or where the subject's mean total daily dose of insulin has not increased by >10% from baseline. If an observation at week 24 is missing or does not meet these criteria, the latest post-baseline value that does will be carried forward (LOCF). The analysis of mean total daily dose of insulin will utilize the latest, non-missing, post-baseline value regardless of rescue. Multiplicity for the primary and secondary endpoints will be controlled via a hierarchical testing procedure that utilizes the full alpha (0.05) for each test. The sequence of testing will be: 1. Change from baseline in HbA1c at Week 24. 2. Change from baseline in PPG AUC at Week 24.3. Change from baseline in 120 minute PPG at Week 24. 4. Proportion of subjects achieving HbA1c <7.0% at Week 24. 5. Change from baseline in FPG to the mean at Week 20 and Week 24. 6. Change from baseline in MTDDI at Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent before participating in the study.
2. Diagnosed with type 2 diabetes.
3. Inadequate glycemic control (screening: HbA1c ≥7.5% and ≤11.0% and FPG<270 mg/dL (15mmol/L). At Day -4 visit, HbA1c ≥7.5% and ≤10.5%. and FPG<270 mg/dL (15mmol/L)).
4. On a stable dose of insulin for 8 weeks or longer prior to screening.
5. If taking metformin, subjects should have been taking the same daily dose for 8 weeks or longer prior to screening.
6. Insulin type should be intermediate-acting or long-acting (basal) or premixed (premixed formulation may include short- or rapid-acting insulin as one component).
7. Body mass index ≤45 kg/m^2.

Exclusion Criteria:

1. Women of childbearing potential unable or unwilling to use acceptable birth control.
2. Women who are pregnant or breastfeeding.
3. Symptoms of poorly controlled diabetes. including but not limited to, marked polyuria and polydipsia with greater than 10% weight loss during the last three months prior to screening or other signs and symptoms.
4. Significant cardiovascular history defined as: myocardial infarction, coronary angioplasty or bypass graft, valvular disease or repair, unstable clinical significant arrhythmia, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident.
5. Congestive heart failure
6. Chronic or repeated intermittent corticosteroid treatment (subjects receiving stable doses of replacement corticosteroid (except dexamethasone) therapy may be enrolled).
7. History of unstable or rapidly progressing renal disease.
8. History of alcohol or drug abuse within the previous year.
9. Unstable major psychiatric disorders.
10. History of hemoglobinopathies
11. Immunocompromised status
12. Severe liver disease.
13. In subjects treated with insulin alone a calculated creatinine clearance <50 ml/min. In patients treated with insulin in combination with metformin a calculated creatinine clearance <60 ml/min or serum creatinine > 1.5 mg/dL in males or > 1.4mg/dL in females.
14. Anemia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Professor, Principal Investigator — People's Hospital of Peking Universty
Locations (11):
- China (11):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Ha'er Bing
  - Research Site, Hefei
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Shiyan

REFERENCES:
- [Result] Drucker DJ. Dipeptidyl peptidase-4 inhibition and the treatment of type 2 diabetes: preclinical biology and mechanisms of action. Diabetes Care. 2007 Jun;30(6):1335-43. doi: 10.2337/dc07-0228. Epub 2007 Mar 2. No abstract available. PMID 17337495
- [Result] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564
- [Result] Fonseca V, Schweizer A, Albrecht D, Baron MA, Chang I, Dejager S. Addition of vildagliptin to insulin improves glycaemic control in type 2 diabetes. Diabetologia. 2007 Jun;50(6):1148-55. doi: 10.1007/s00125-007-0633-0. Epub 2007 Mar 27. PMID 17387446
- [Result] Pan CY, Yang W, Tou C, Gause-Nilsson I, Zhao J. Efficacy and safety of saxagliptin in drug-naive Asian patients with type 2 diabetes mellitus: a randomized controlled trial. Diabetes Metab Res Rev. 2012 Mar;28(3):268-75. doi: 10.1002/dmrr.1306. PMID 22081481
- [Result] Vilsboll T, Rosenstock J, Yki-Jarvinen H, Cefalu WT, Chen Y, Luo E, Musser B, Andryuk PJ, Ling Y, Kaufman KD, Amatruda JM, Engel SS, Katz L. Efficacy and safety of sitagliptin when added to insulin therapy in patients with type 2 diabetes. Diabetes Obes Metab. 2010 Feb;12(2):167-77. doi: 10.1111/j.1463-1326.2009.01173.x. PMID 20092585
- [Result] Yang W, Pan CY, Tou C, Zhao J, Gause-Nilsson I. Efficacy and safety of saxagliptin added to metformin in Asian people with type 2 diabetes mellitus: a randomized controlled trial. Diabetes Res Clin Pract. 2011 Nov;94(2):217-24. doi: 10.1016/j.diabres.2011.07.035. Epub 2011 Aug 26. PMID 21871686
- [Derived] Chen Y, Liu X, Li Q, Ma J, Lv X, Guo L, Wang C, Shi Y, Li Y, Johnsson E, Wang M, Zhao J, Ji L. Saxagliptin add-on therapy in Chinese patients with type 2 diabetes inadequately controlled by insulin with or without metformin: Results from the SUPER study, a randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2018 Apr;20(4):1044-1049. doi: 10.1111/dom.13161. Epub 2017 Dec 18. PMID 29144061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 22 sites in the People's Republic of China (PRC).The first patient was enrolled on 07 May 2014 and the last patient completed the study on 26 February 2016. The study was divided into a single-blind placebo lead-in period of 8 weeks, a treatment period of 24 weeks and a follow-up phase of 4 weeks.
Pre-assignment Details: 953 patients were enrolled, of which 641 patients took at least 1 dose of study drug and entered the lead-in period. A total of 312 patients did not enter the lead-in period (289 did not fulfill eligibility criteria, 21 due to subject decision, 1 each for severe non-compliance to protocol and other reasons) and 466 patients were randomized.
Groups:
- Saxagliptin Plus Insulin: Saxagliptin 5 mg plus insulin
- Vs. Placebo Plus Insulin: Patients receiving placebo 5 mg plus insulin
Period: Overall Study
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Started | 234 (Number of patients who were randomized) | 232 (Number of patients who were randomized)
Completed | 218 (Number of patients who completed 24 weeks of treatment) | 213 (Of the 19 who did not complete, 1 did not take study medication after randomization.)
Not Completed | 16 | 19
Not completed — Did not take study medication | 0 | 1
Not completed — Study specific discontinuation criteria | 6 | 1
Not completed — Other listed | 2 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 4 | 3
Not completed — Withdrawal by Subject | 4 | 12

BASELINE CHARACTERISTICS:
Population: Note that 462 indicates the number of patients in the Full Analysis set (out of 466 randomized, 1 did not take study drug and 3 did not have 1 baseline or post baseline efficacy assessment).
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin | Total
Number analyzed (Participants) | 232 | 230 | 462
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.3 (7.93) | 58.9 (8.17) | 59.1 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 130 | 253
  Male | 109 | 100 | 209
Baseline HbA1C [Mean (Standard Deviation); unit: %] | 8.52 (0.69) | 8.53 (0.70) | 8.53 (0.69)
Duration of diabetes [Mean (Standard Deviation); unit: Years] | 13.4 (7.28) | 13.3 (6.35) | 13.4 (6.83)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 167.94 (31.39) | 167.34 (32.86) | 167.64 (32.10)
0-180 min Post Prandial Glucose AUC [Mean (Standard Deviation); unit: mg*min/dL] | 45457.6 (8433.08) | 43851.4 (9051.26) | 44661.5 (8772.22)
120-min Post Prandial Glucose [Mean (Standard Deviation); unit: mg/dL] | 278.0 (58.00) | 270.0 (63.30) | 274.0 (60.76)
Fasting Glucagon [Mean (Standard Deviation); unit: pg/dL] | 40.007 (23.68) | 40.231 (21.06) | 40.119 (22.39)
Fasting C-peptide [Mean (Standard Deviation); unit: ng/dL] | 1.029 (0.52) | 1.012 (0.58) | 1.020 (0.55)
Metformin use at enrolment [Number; unit: Participants]
  Yes | 155 | 154 | 309
  No | 77 | 76 | 153
Mean Tolerated Daily Dose of Insulin [Mean (Standard Deviation); unit: Insulin Dose Units] | 38.6 (16.49) | 38.9 (14.68) | 38.7 (15.60)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Time Frame: Baseline to 24 weeks
Population: 229 and 227 indicate the number of participants with non-missing baseline and Week 24 values in the Full Analysis Set of 232 and 230 respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 229 | 227
Percentage change | -0.64 [-0.74 to -0.55] | -0.06 [-0.16 to 0.04]
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -0.58, 95% CI 2-sided [-0.72 to -0.45], Standard Error of Mean 0.07

2. Secondary Outcome: Change in Postprandial Glucose AUC From Baseline to Week 24 During a Meal Tolerance Test
Time Frame: Baseline to 24 weeks
Population: 213 and 206 indicate the number of participants with non-missing baseline and Week 24 values in the Full Analysis Set of 232 and 230 respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg*min/dL
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 213 | 206
mg*min/dL | -4702.2 [-5813.3 to -3591.0] | 1431.0 [294.4 to 2567.7]
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -6133.2, 95% CI 2-sided [-7668.5 to -4597.9], Standard Error of Mean 781.06

3. Secondary Outcome: Analysis of Change in 120-minute PPG From Baseline to Week 24 During a Meal Tolerance Test
Time Frame: Baseline to 24 weeks
Population: 215 and 211 indicate the number of participants with non-missing baseline and Week 24 values in the Full Analysis Set of 232 and 230 respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 215 | 211
mg/dL | -30.28 [-37.76 to -22.80] | 8.84 [1.25 to 16.42]
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least squares mean = -39.11, 95% CI 2-sided [-49.41 to -28.82], Standard Error of Mean 5.24

4. Secondary Outcome: Percentage of Patients Achieving a Therapeutic Glycaemic Response of HbA1c <7%
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number; unit: % of participants
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 229 | 227
% of participants | 11.4 | 3.5
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p = 0.002, Difference in proportions; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [3.1 to 12.6]

5. Secondary Outcome: The Analysis of Change in Fasting Plasma Glucose From Baseline to Week 24 (This Was the Average of Weeks 20 and 24)
Time Frame: Baseline to Average of Weeks 20 and 24
Population: 232 and 229 indicate the number of participants with non-missing baseline and Week 24 values in the Full Analysis Set of 232 and 229 for this outcome measure respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 232 | 229
mg/dL | -11.23 [-15.34 to -7.11] | 4.65 [0.50 to 8.80]
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -15.88, 95% CI 2-sided [-21.53 to -10.22], Standard Error of Mean 2.88

6. Secondary Outcome: Analysis of Change in Mean Total Daily Dose of Insulin From Baseline to Week 24
Time Frame: Baseline to 24 weeks
Population: 232 and 230 indicate the number of participants with non-missing baseline and Week 24 values in the Full Analysis Set of 232 and 230 respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: IU
Arm/Group | Saxagliptin Plus Insulin | Vs. Placebo Plus Insulin
Number analyzed (Participants) | 232 | 230
IU | -0.09 [-0.32 to 0.14] | 0.04 [-0.19 to 0.27]
Statistical Analysis 1: Comparison: Vs. Placebo Plus Insulin; Test type: Superiority or Other; p = 0.430, ANCOVA; Difference in Least squares mean = -0.13, 95% CI 2-sided [-0.44 to 0.19], Standard Error of Mean 0.16

ADVERSE EVENTS:
Description: Total numbers at risk indicate the number of participants in the Safety Analysis set. Out of 466 randomized, 1 did not take study drug.
Arm/Group | PLACEBO QD + INSULIN WITH OR WITHOUT METFORMIN | SAXAGLIPTIN 5 MG QD + INSULIN WITH OR WITHOUT METFORMIN
Serious Adverse Events (participants affected / at risk) | 14/231 | 12/234
Other Adverse Events (participants affected / at risk) | 96/231 | 89/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO QD + INSULIN WITH OR WITHOUT METFORMIN (N=231) | SAXAGLIPTIN 5 MG QD + INSULIN WITH OR WITHOUT METFORMIN (N=234)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO QD + INSULIN WITH OR WITHOUT METFORMIN (N=231) | SAXAGLIPTIN 5 MG QD + INSULIN WITH OR WITHOUT METFORMIN (N=234)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysbacteriosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 5 (5)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 3 (4)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (12) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2) | 6 (6)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 2 (3)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 55 (131) | 51 (171)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without limitation to any other right of AstraZeneca hereunder, Institution and Principal Investigator acknowledge and agree that only AZ as Sponsor will register the Study and post the Study results in accordance with AZ internal policy on one or more publicly-accessible trial registries and websites (including the publicly-funded website http://www.clinicaltrials.gov/ and on its own website http://www.astrazenecaclinicaltrials.com) to avoid duplication.